CLINICAL TRIAL: NCT01804517
Title: Impact of a Nursing Intervention on the Clinical Evolution of Patients at a University Migraine Clinic
Brief Title: Impact of a Nurse for Migraine Management: the IMPACT Project
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Notre-Dame Hospital, Montreal, Quebec, Canada (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Elizabeth Leroux, M.D. Neurologist, FRCPC, Notre-Dame Hospital, Montreal, Quebec, Canada
Other Study IDs: IMPACT
Record Dates: First submitted 2013-02-23; First posted 2013-03-05 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Migraine Without Aura; Migraine With Aura; Chronic Migraine
Keywords: migraine
MeSH Terms: conditions — Migraine without Aura; Migraine with Aura; Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Physician based approach: Patients will be managed as usual at the clinic without the intervention of the nurse.
- Physician and nurse: Patients will be managed with the help of the nurse for education and follow-up.

SUMMARY:
Headache disorders are prevalent, disabling, under recognized, under diagnosed and under treated. Migraine has a prevalence of 10% in men and 25% in women in Canada. The treatment of migraine is based on patient education (lifestyle habit modification, trigger avoidance), and pharmacological acute treatment and prophylaxis. A multidisciplinary approach allows a repartition of tasks between different health professionals.

In a 2010 meeting, the Canadian Headache Society members supported the concept of Headache Centers, and a headache nurse was judged as an essential component of such centers.

Gaul has reviewed the structured multidisciplinary approach that could be used in a headache centre and the existing studies using such structures. Five studies did include a headache nurse. No study did observe the impact of a nurse only. Resources in medical care are limited. One study did use a program of 96 hours, which does not seem realistic on the long-term and for a large pool of patients in a public hospital. Patients are not always able to pay for paramedical help such as physiotherapy and psychotherapy. Even if they do, finding a specialized therapist for chronic headache is difficult. Defining the role of a nurse and demonstrating the impact on patient care is therefore a first step in the concept of a headache center. Possible roles of a headache nurse according to Gaul are patient education, follow-up of the treatment plan, addressing patient queries, and monitoring of patient progress. The headache nurse may also participate in research projects. In a hospital Headache Clinic, the nurse may be involved in intra-venous treatments and blood sampling for research.

In summary, evidence to demonstrate the impact of a nurse in a headache clinic is lacking. We propose to study this aspect prospectively. A study with positive findings would encourage health ministers to fund and support headache nurses for headache centers across Canada for headache management. Chronic headache and therefore chronic migraine would be a focus of such centers, since most patients seen in specialized centers are chronic.

HYPOTHESIS: The addition of a headache nurse to the headache team will help the CHUM Migraine Clinic to improve treatment outcome, and reduce the burden of headache. This multidisciplinary approach will also allow a higher efficiency of the team.

DETAILED DESCRIPTION:
STUDY DESIGN:

The goal of this study is to compare two treatment approaches for migraineurs. The first approach will be based on the physician only and is limited to fixed appointments (control group). The second approach will be based on a team involving a headache nurse (active group) who will participate in patient education and follow-up. The goal is to improve patient outcome but also physician productivity.

First 100 patients (control group, phase 1): patients with episodic and chronic migraine will be screened, sign consent and be enrolled. They will be seen by the physician only, without the nurse's support. This situation will reproduce the actual conditions at the clinic. During this phase, the nurse will be involved in the follow-up of known patients (who will not be included in the protocol) and data collection. She will develop her headache management abilities and help the physicians to develop some educational tools for patients.

Following 100 patients (active group, phase 2) : patients with episodic and chronic migraine will be screened and enroled. They will be seen by the physician and nurse team, with a treatment plan tailored to specific needs including regular scheduled visits, follow-up of chronification factors and educational sessions. Phone call follow-ups will be planned. Patients will have an easier and quicker contact with the team in an emergency situation.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18 or more
* Diagnosis of migraine, chronic or episodic, at the first visit. We expect the majority of patients to suffer form frequent or chronic migraine.
* Consent to participate in the CHUM Migraine Clinic IMPACT project.
* For future post-hoc analysis, groups will be stratified according to baseline headache frequency (all severity included), assessed retrospectively at the first visit:

  * <6 headache days per month,
  * 6 to 14 headache days per month
  * 15 or more headache days per month

EXCLUSION CRITERIA:

* Patients whom first headache diagnosis is not migraine (for example post-traumatic headache, cluster headache, trigeminal neuralgia, facial pain).
* Women with ongoing or planned pregnancy.
* Patient with an active psychiatric condition (needing hospitalisation or psychosis).
* Patient with mental retardation impairing assessment or follow-up.
* Patient with an active medical condition which may lead to frequent hospitalisations (eg active cancer, organ graft, hemodialysis etc). This will be determined and detailed by the evaluating physician.
* Active drug addiction or alcoholism.
* Active follow-up at a pain clinic.
* Patient speaking a language other than french and incapable to communicate in a reliable way.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at the migraine clinic at the Notre-Dame Hospital in Montreal
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Hit-6 score change | Baseline and 8 months
  HIT-6 score change between inclusion and 8 month.

SECONDARY OUTCOMES:
Frequency of moderate and severe headache days | Baseline and 8 months
  Variation in the frequency of moderate or severe headache days per month between the first, fourth and eighth month after inclusion.
Frequency of headache days | Baseline and 8 months
  Change in the frequency of headache days, all severity included, between the first month and the seventh and eight months following inclusion.
Chronic headache status | Baseline and 1 year
  Percent of patients who were chronic (more than 3 months with >15 headache days per month, retrospective) at entry and were episodic at one year (according to calendars).
Medication overuse | Baseline and 8 months
  Percent of patients with medication overuse at entry and were not overusing anymore at 8 months.
Acute medication intake | Baseline and 8 months
  Change in the number of days per month with acute medication use between the first month after inclusion and the seventh and eight months following inclusion.
Efficacy of acute treatment | at 8 months
  Percent of patients who succeeded in finding a successful and properly used acute treatment at month eight, according to four criteria: efficacy, reliability, absence of recurrence, absence of significant side effects.
Response rate to prophylactics | at 8 months
  Percent of patients who did complete a successful (>50% response and no significant side-effects) preventive treatment trial at month eight after inclusion.
Short Form 12 score | Baseline and 8 months
  Change in SF-12 scores between inclusion and third visit. SF-12 is a quality of life questionnaire.
Visits to the emergency department | over 1 year
  Number of headache-related emergency department visits per patient during the year following their inclusion.
Severe adverse effects from treatments | over 1 year
  Percent of patients with a severe adverse effect from a treatment (necessitating hospitalization, emergency visit or specific treatment).
Phone calls returned | per 1 month
  Number of phone calls returned per month
Patient satisfaction | at 8 months
  Satisfaction of patients, evaluated by a customized questionnaire.
Phone call return delay | for each phone call, mean
  Mean delay for returning the call (number of week days between the date of the call and the date of the return).
Global improvement | at 8 months
  Evaluation of physician of the global improvement of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Leroux, M.D., Principal Investigator — FRCPC
Locations (1):
- Hôpital Notre-Dame, Montreal, Quebec, Canada